CLINICAL TRIAL: NCT02647853
Title: A Randomized, Placebo-controlled, Double-blind, Multiple-ascending-dose, Phase 1 Study to Assess the Safety and Tolerability of TAT4 Gel
Brief Title: Phase 1 Study to Assess the Safety and Tolerability of TAT4 Gel in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Topokine Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAT4 A1
Record Dates: First submitted 2016-01-03; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Nasolabial Folds; Lipoatrophy; Lipodystrophy
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAT4 Gel concentration A (Experimental): TAT4 Gel concentration A applied once daily to 50 cm2 for 14 days.
  Interventions: Drug: TAT4 Gel concentration A
- TAT4 Gel concentration B (Experimental): TAT4 Gel concentration B applied once daily to 50 cm2 for 14 days.
  Interventions: Drug: TAT4 Gel concentration B
- Placebo (Placebo Comparator): Placebo product once daily to 50 cm2 for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAT4 Gel concentration A
  Arms: TAT4 Gel concentration A
Drug: TAT4 Gel concentration B
  Arms: TAT4 Gel concentration B
Drug: Placebo
  Arms: Placebo

SUMMARY:
This Phase 1, randomized, placebo-controlled, double-blind, healthy volunteer study tested the safety, tolerability, and plasma pharmacokinetics of two different concentrations of TAT4 Gel administered once daily to 50 cm2 of skin for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 40-70 years old
* Healthy volunteers
* Provision of informed consent

Exclusion Criteria:

* History of skin hypersensitivity
* Abnormality on screening assessments

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Adverse Event rates | 21 days
  Adverse event rates by System Organ Class, as graded by current CTCAE

SECONDARY OUTCOMES:
Plasma pharmacokinetics (Cmax) | Days 1 and 13
Plasma pharmacokinetics (Tmax) | Days 1 and 13
Plasma pharmacokinetics (AUC0-24) | Day 1 and 13

CONTACTS AND LOCATIONS:
Locations (1):
- Topokine Clinical Site, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No